CLINICAL TRIAL: NCT00002967
Title: A Clinical Trial to Evaluate the Benefit of Adding Octreotide (SMS 201-995 PA LAR) to Tamoxifen Alone or to Tamoxifen and Chemotherapy in Patients With Axillary Node-Negative, Estrogen-Receptor-Positive, Primary Invasive Breast Cancer
Brief Title: Octreotide, Tamoxifen, and Chemotherapy in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065472; NSABP-B-29
Record Dates: First submitted 1999-11-01; First posted 2004-09-03 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; invasive ductal breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast | interventions — Cyclophosphamide; Doxorubicin; Tamoxifen

INTERVENTIONS:
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: octreotide pamoate
Drug: tamoxifen citrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining hormone therapy with chemotherapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to study the effectiveness of tamoxifen, octreotide, and chemotherapy in treating women who have stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether the addition of octreotide pamoate to tamoxifen alone or to tamoxifen and chemotherapy improves the disease free survival of patients with primary invasive breast cancer with estrogen receptor (ER) positive tumors and histologically negative axillary lymph nodes or histologically negative sentinel lymph nodes if participating in NSABP B-32. II. Determine whether the rate of endometrial cancer associated with tamoxifen is altered by the concurrent administration of octreotide pamoate. III. Determine whether the addition of octreotide pamoate to tamoxifen decreases the rate of opposite breast cancer more than tamoxifen alone. IV. Evaluate the incidence of gallstone formation (including the development of symptoms and complications of biliary tract disease), hyper and hypoglycemia, hypothyroidism, and vitamin B12 deficiency in patients treated with octreotide pamoate in comparison with patients not treated with octreotide pamoate.

OUTLINE: This is a randomized study. Patients are randomized into one of four treatment arms. Arm I: Patients receive oral tamoxifen (TMX) daily continously for 5 years. Lumpectomy patients receive breast radiotherapy following recovery from surgery. Arm II: Patients receive TMX as in Arm I and octreotide pamoate (SMS 201-995 pa LAR) intramuscularly (IM) every 21 days for 4 doses, followed by octreotide pamoate IM for 28 days for 23 additional doses. Lumpectomy patients receive breast radiotherapy following recovery from surgery. Arm III: Patients receive doxorubicin (DOX) IV and cyclophosphamide (CTX) IV every 3 weeks for 4 courses and TMX as in Arm I. Lumpectomy patients receive breast radiotherapy after recovery from chemotherapy. Arm IV: Patients receive DOX and CTX as in Arm III, TMX as in Arm I, and octreotide pamoate as in Arm II. Patients receive TMX and octreotide pamoate on day 1 of first course of chemotherapy. Lumpectomy patients receive breast radiotherapy after recovery from chemotherapy.

PROJECTED ACCRUAL: Total accrual of 3,000 patients will be acrrued for this study over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed Stage I, IIA or IIB invasive adenocarcinoma of the breast with T1-3, pN0 and M0 classification Must have undergone total mastectomy or lumpectomy followed by an axillary dissection or sentinel node resection if participating in NSABP B-32 Histologically negative axillary lymph nodes OR Histologically negative sentinel lymph nodes if participating in NSABP B-32 Lumpectomy and axillary dissection acceptable only if margins of resected specimen are histologically free of invasive tumor or ductal carcinoma in situ and other dominant masses within the ipsilateral breast remnant are histologically confirmed to be benign Additional operation after resection is allowed in order to obtain clear margins No bilateral malignancy of the breast ER positive tumors as defined by at least one of the following: At least 10 fmol/mg cytosol protein by either dextran-coated charcoal or sucrose density gradient methods Positive or not definitely negative results by the enzyme immunoassay method (EIA) or by immunocytochemical assay No more than 63 days from time of initial cytologic or histologic diagnosis of breast cancer till randomization No bone metastases (confirmation must be made for those with skeletal pain) Tumor must be no greater than 5 cm in its greatest dimension for patients who are treated by lumpectomy and axillary dissection Hormone receptor status: Estrogen receptor positive

PATIENT CHARACTERISTICS: Age: Not specified Sex: Female Menopausal status: Not specified Life expectancy: At least 10 years (excluding diagnosis of cancer) Performance status: Not specified Hematopoietic: WBC at least 4,000/mm3 Platelet count postoperative at least 100,000/mm3 Hepatic: Bilirubin normal SGOT/SGPT normal Renal: Creatinine normal Cardiovascular: No cardiac disease that would preclude the use of doxorubicin (for patients who are to receive adjuvant chemotherapy in this study), including: Myocardial infarction Angina pectoris that requires antianginal medication History of congestive heart failure Arrhythmia associated with concurrent heart failure or cardiac dysfunction Valvular disease with cardiac compromise Cardiomegaly or ventricular hypertrophy unless left ventricular function is within normal limits Poorly controlled hypertension Other: No prior invasive breast cancer or ductal carcimoma in situ No systemic disease that would preclude patients from any part of study No history of symptomatic gallbladder or biliary tract disease unless patient has undergone cholecystectomy No ulceration, erythema, infiltration of the skin or underlying chest wall (complete fixation), peau d'orange, or skin edema of any magnitude No prior nonbreast malignancies in past 10 years except: Squamous or basal cell carcinoma of the skin that has been effectively treated Carcinoma in situ of the cervix that has been treated by operation only Lobular carcinoma in situ of the ipsilateral or contralateral breast treated by segmented resection only No psychiatric or addictive disorders Not pregnant or nursing Negative pregnancy test

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy for breast cancer Chemotherapy: No prior chemotherapy for breast cancer No prior anthracycline therapy for patients who are to receive adjuvant chemotherapy in this study Endocrine therapy: No prior endocrine therapy for breast cancer Must discontinue any sex hormonal therapy before prior to and during study Radiotherapy: No prior radiotherapy for breast cancer No breast radiation therapy before randomization for patients who receive lumpectomy Surgery: See Disease Characteristics At least 2 weeks since last surgical procedure Other: No concurrent cyclosporine therapy No concurrent heparin or warfarin anticoagulation therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-05; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard G. Margolese, MD, Study Chair — Jewish General Hospital
Locations (108):
- United States (106):
  - Baptist Medical Center - Birmingham, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Scripps Clinic and Research Foundation - La Jolla, La Jolla, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Sutter Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Ocala Oncology Center, Ocala, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Winship Cancer Center, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Illinois Masonic Medical Center, Chicago, Illinois
  - Highland Park Hospital, Highland Park, Illinois
  - West Suburban Hospital Medical Center, Oak Park, Illinois
  - Rockford Clinic, Rockford, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Methodist Cancer Center - Indianapolis, Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Lucille Parker Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - Norton Healthcare System, Louisville, Kentucky
  - Louisiana State University Medical Center - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Franklin Square Hospital Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic - Burlington, Burlington, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - St. Louis University School of Medicine, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Albany Regional Cancer Center, Albany, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Genesee Hospital - Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Akron City Hospital, Akron, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Jewish Hospital of Cincinnati, Inc., Cincinnati, Ohio
  - Meridia South Pointe Hospital, Cleveland, Ohio
  - Mount Sinai Medical Center - Cleveland, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - St. Francis Hospital/Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - St. Luke's Network - Bethlehem, Bethlehem, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Kent County Memorial Hospital - Rhode Island, Warwick, Rhode Island
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Virginia Oncology Associates, Newport News, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec

REFERENCES:
- [Background] Chapman JA, Costantino JP, Dong B, et al.: Randomized trials of adjuvant tamoxifen versus tamoxifen and octreotide LAR in early-stage breast cancer: NCIC CTG MA.14 and NSABP B-29. [Abstract] J Clin Oncol 30 (Suppl 15): A-538, 2012.
- [Background] Soran A, Nesbitt L, Mamounas EP, Lembersky B, Bryant J, Anderson S, Brown A, Passarello M. Centralized medical monitoring in phase III clinical trials: the National Surgical Adjuvant Breast and Bowel Project (NSABP) experience. Clin Trials. 2006;3(5):478-85. doi: 10.1177/1740774506070747. PMID 17060221
- [Derived] Chapman JA, Costantino JP, Dong B, Margolese RG, Pritchard KI, Shepherd LE, Gelmon KA, Wolmark N, Pollak MN. Octreotide LAR and tamoxifen versus tamoxifen in phase III randomize early breast cancer trials: NCIC CTG MA.14 and NSABP B-29. Breast Cancer Res Treat. 2015 Sep;153(2):353-60. doi: 10.1007/s10549-015-3547-4. Epub 2015 Aug 15. PMID 26276354